CLINICAL TRIAL: NCT03817177
Title: Seoul National University Hospital Department of Anesthesiology and Pain Medicine
Brief Title: Application of High Flow Nasal Cannula for Prevention of Post-extubation Atelectasis in Children Undergoing Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, principle investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1812-111-998
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal prong (Placebo Comparator): conventional nasal prong application after the surgery in postanesthetic care unit (PACU)
  Interventions: Procedure: nasal prong
- high flow nasal cannula oxygenation (Experimental): high flow nasal cannula application after the surgery in postanesthetic care unit (PACU)
  Interventions: Procedure: high flow nasal cannula oxygenation

INTERVENTIONS:
Procedure: high flow nasal cannula oxygenation — high flow nasal cannula application in PACU
  Arms: high flow nasal cannula oxygenation
Procedure: nasal prong — conventional nasal prong application in PACU
  Arms: nasal prong

SUMMARY:
postoperative atelectasis observation by ultrasound after application of high flow nasal cannula oxygenation

DETAILED DESCRIPTION:
After surgery, postoperative atelectasis observation by ultrasound grading comparison between application of conventional nasal prong and high flow nasal cannula device

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia

Exclusion Criteria:

* preterm
* bronchopulmonary dysplasia
* upper respiratory infection history
* respiratory disease
* cardiac surgery

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-03-02 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
lung sound score | 30 minutes after arrival of postanesthetic care unit
  0: Normal aeration (N): presence of lung sliding with A lines or fewer than two isolated B lines
  1. Moderate loss of lung aeration: multiple well-defined B lines (B1 lines)
  2. Severe loss of lung aeration: multiple coalescent B lines (B2 lines)
  3. Lung consolidation (C): the presence of a tissue pattern characterized by dynamic air

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JH, Ji SH, Jang YE, Kim EH, Kim JT, Kim HS. Application of a High-Flow Nasal Cannula for Prevention of Postextubation Atelectasis in Children Undergoing Surgery: A Randomized Controlled Trial. Anesth Analg. 2021 Aug 1;133(2):474-482. doi: 10.1213/ANE.0000000000005285. PMID 33181560